CLINICAL TRIAL: NCT01308177
Title: Efficacy of an Ecabet Sodium and Proton Pump Inhibitor (PPI) Combination Therapy in the Treatment of Iatrogenic Ulcer After Endoscopic Submucosal Dissection: A Prospective Randomized Controlled Trial
Brief Title: Efficacy of Ecabet Sodium and Proton Pump Inhibitor Combination Therapy in the Treatment of Iatrogenic Ulcer After Endoscopic Submucosal Dissection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Samsung Medical Center (Other)
Responsible Party: Jaej Kim, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-10-044
Record Dates: First submitted 2011-03-02; First posted 2011-03-03 (Estimated); Last update posted 2011-03-03 (Estimated); Status verified 2011-03

CONDITIONS: Delayed Bleeding,; Healing Ulcer; Quality of Ulcer
MeSH Terms: interventions — ecabet

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- PPI+placebo (Placebo Comparator)
  Interventions: Drug: Ecabet
- PPI+ES (Active Comparator)
  Interventions: Drug: Ecabet

INTERVENTIONS:
Drug: Ecabet — comparison between PPI+ ES (lanston 30mg bid+ ES 1g/1.5g/pkg bid) and PPI+placebo (lanston 30mg bid)for 28 days

SUMMARY:
* Endoscopic submucosal dissection (ESD) is widely indicated to treat gastric adenomas and early gastric cancer (EGC).ESD is able to obtain en bloc resection of larger specimens. However, ESD has more frequent complications (delayed bleeding, ulcer healing, ulcer pain, and etc) due to a more complex procedure. To prevent delayed bleeding, to induce rapid ulcer healing, and to control the ulcer pain acid-suppressing agents (PPI, H2RA) are generally administered. although PPIs are widely indicated as first-line drugs for peptic ulcers, PPI drugs are not fully superior to H2RAs or other combination drugs for treatment of iatrogenic ulcer healing and delayed bleeding.
* Ecabet sodium (ES)is a widely used mucoprotective agent for the treatment of gastric ulcers. Recently, one study showed the additional benefits of using ES in combination with the PPI after ESD. however, this study did not show the difference of delayed bleeding and the benefit of ulcer pain control. thus, our study prospectively evaluated the difference of delayed bleeding and the benefit of ulcer pain control after ESD.

ELIGIBILITY:
Inclusion Criteria:

* gastric adenomas or differentiated EGC (any size without ulcers or signs of submucosal invasion; intramucosal differentiated-type EGC < 3 cm with a scar; and no lymph node involvement or metastasis by CT)

Exclusion Criteria:

* recent use of a PPI, H2RA, bismuth, and antibiotics
* current use of aspirin, non-steroidal anti-inflammatory drugs, or corticosteroids
* Helicobacter pylori infection not evaluated appropriately by endoscopic biopsy and serology
* a history of subtotal gastrectomy; patients who underwent surgery due to ESD complications; known hypersensitivity to PPIs
* chronic co-morbid disease, such as chronic liver and renal disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
to determine the difference in delayed bleeding with PPI or PPI+ES | the time of bleeding occured or post 4 weeks after ESD

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea